CLINICAL TRIAL: NCT03649321
Title: A phase1b/2 Clinical Trial of Chemotherapy and the AXL-inhibitor Bemcentinib for Patients With Metastatic Pancreatic Cancer
Brief Title: Clinical Trial of Chemotherapy and Bemcentinib for Metastatic Pancreatic Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Funding was terminated early because research interests were going in a different direction.
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Triligent International (Industry); Translational Genomics Research Institute (Other); BerGenBio ASA (Industry)
Responsible Party: Principal Investigator, Syed Kazmi, Associate Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 062018-024
Record Dates: First submitted 2018-08-16; First posted 2018-08-28 (Actual); Results first posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-10

CONDITIONS: Cancer of Pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — bemcentinib; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Paclitaxel; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1b (Experimental): bemcentinib 200 mg oral daily every 21 days. Nab-paclitaxel 100 mg/m^2 Day 1 /8 every 21 days. Gemcitabine 800 mg/m^2 Day 1 /8 every 21 days. Cisplatin 25 mg/m^2 Day 1 /8 every 21 days.
  Interventions: Drug: Bemcentinib; Drug: Nab-paclitaxel; Drug: Gemcitabine; Drug: Cisplatin
- Phase 2 (Experimental): bemcentinib 200 mg oral daily every 28 days. Nab-paclitaxel 125 mg/m^2 Day 1 /8 /15 every 28 days. Gemcitabine 1000 mg/m^2 Day 1 /8 /15 every 28 days.
  Interventions: Drug: Bemcentinib; Drug: Nab-paclitaxel; Drug: Gemcitabine

INTERVENTIONS:
Drug: Bemcentinib — 200mg orally starting Cycle 1 day 2 every 21 days or 28 days.
Drug: Nab-paclitaxel — 25 mg/m^2 Day 1 /8 every 21 days or 28 days.
  Other Names: ABI-007, PACLITAXEL
Drug: Gemcitabine — Gemcitabine 1000 mg/m^2 Day 1 /8 every 21 days or 28 days
  Other Names: GemzarTM
Drug: Cisplatin — Cisplatin 25 mg/m^2 Day 1 /8 every 21 days
  Arms: Phase 1b

SUMMARY:
Determine the overall response rate (ORR) of bemcentinib plus chemotherapy (nab-paclitaxel/gemcitabine) in patients with metastatic pancreatic adenocarcinoma.

DETAILED DESCRIPTION:
Bemcentinib inhibits pancreatic cancer proliferation as monotherapy and in combination with gemcitabine through inhibition of the Axl pathway. The combination of nab-paclitaxel/gemcitabine has encouraging signs of clinical activity in patients with metastatic pancreatic cancer38. We would like to build on this combination in a biomarker driven phase 1b/2 clinical trial of bemcentinib in nab-paclitaxel/gemcitabine for patients with metastatic pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and the willingness to sign a written informed consent.
2. Patients must have histologically or cytologically confirmed recurrent or metastatic pancreatic adenocarcinoma.
3. No prior systemic therapy for metastatic or recurrent disease.

   * Prior adjuvant therapy, if completed more than 6 months prior to date of enrollment, is acceptable.
   * Radiosensitizing chemotherapy, if completed at least 4 weeks from date of enrollment, is acceptable.
4. Measurable disease per RECIST1.1 criteria
5. Age 18-70 years at the time of enrollment
6. ECOG performance status 0 or 1
7. Have resolution of toxic effect(s) or intervention complication to Grade 1 or less (except alopecia) from any prior chemotherapy, major surgery, or radiation therapy of >30 Gy.
8. Adequate hematologic, hepatic, and renal function. All screening labs should be performed within 14 days of enrollment date.

   * Hemoglobin ≥ 10 g/dL
   * ANC ≥ 1,500/µL
   * Platelets ≥ 100,000/µL
   * Total bilirubin < 1.5 x institutional ULN
   * AST (SGOT) & ALT(SGPT)≤ 2.5 x institutional ULN in patients without known liver metastasis; ≤ 5 x institutional ULN in patients with known liver metastasis
   * Serum creatinine ≤ 1.5 times ULN, and calculated creatinine clearance ≥ 60 mL/min using the Cockcroft-Gault equation)
   * INR or PT International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5 times the ULN
   * Albumin ≥ 3.0 g/dL
9. Female patients of childbearing potential must have a negative pregnancy test (either urine or serum pregnancy test). If the urine pregnancy test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

   * Has not undergone a hysterectomy or bilateral oophorectomy; or
   * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
10. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 120 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician, or study team member, immediately.

Exclusion Criteria:

1. Is currently participating and receiving study therapy in a first line setting for metastatic or recurrent pancreatic adenocarcinoma.
2. Participated in a study of an investigational agent or used an investigational device within 4 weeks of the first dose of study treatment.
3. Patients with known untreated brain metastases. Patients without known or suspected brain metastases do not require radiologic imaging prior to enrollment.
4. Has a known additional malignancy that is progressing or requires active treatment. Note: Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
5. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, significant pulmonary disease (shortness of breath at rest or mild exertion), or uncontrolled infection or psychiatric illness/social situations that would limit compliance with study requirements.
6. History of the following cardiac conditions:
7. Congestive cardiac failure of >Grade II severity according to the NYHA (defined as symptomatic at less than ordinary levels of activity);
8. Ischemic cardiac event including myocardial infarction within 3 months prior to date of enrollment
9. Uncontrolled cardiac disease, including unstable angina pectoris, uncontrolled hypertension (i.e. sustained systolic BP >160 mmHg or diastolic BP >90 mmHg), cardiac arrhythmia, or need to change medication due to lack of disease control within 6 weeks prior to date of enrollment;
10. History or presence of sustained bradycardia (≤55 BPM), left bundle branch block, cardiac pacemaker or ventricular arrhythmia. Note: Patients with a supraventricular arrhythmia requiring medical treatment, but with a normal ventricular rate are eligible;
11. Known family history or personal history of long QTc syndrome or previous drug-induced QTc prolongation of at least Grade 3 (QTc >500 ms).
12. Abnormal left ventricular ejection fraction (LVEF) on ECHO or MUGA less than <45%.
13. Current treatment with any agent known to cause Torsades de Pointes which cannot be discontinued at least five half-lives or two weeks prior to the first dose of study treatment.
14. Screening 12-lead ECG, in triplicate, with a measurable QTc interval according to Fridericia's correction >450 ms.
15. Known active infection with human immunodeficiency virus (HIV), hepatitis B or C viruses (screening not required, follow institutional practice):
16. Patients who have a history of hepatitis B infection are eligible provided they are hepatitis B surface antigen negative.
17. Patients who have a history of hepatitis C infection are eligible provided they have no evidence of hepatitis C ribonucleic acid using a quantitative polymerase chain reaction assay at least 6 months after completing treatment for hepatitis C infection.
18. Active, clinically significant serious infection requiring treatment with antibiotics, anti-virals or anti-fungals.
19. Treatment with any medication which is predominantly metabolized by CYP3A4 and has a narrow therapeutic index
20. Major surgery within 4 weeks prior to date of enrollment; excluding skin biopsies and procedures for insertion of central venous access devices.
21. Inability to tolerate oral medication
22. Existing gastrointestinal disease affecting drug absorption such as celiac disease or Crohn's disease, or previous bowel resection which is considered to be clinically significant or could interfere with absorption.
23. Known lactose intolerance
24. Is pregnant or breastfeeding
25. Any significant medical condition lab abnormality, or psychiatric illness, in the opinion of the investigator, that might interfere with the patient's participation in the study or in the evaluation of the study results.
26. Unwillingness or inability to comply with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2022-06-27 (Actual); Study Completion 2022-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Syed Kazmi, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Phase 1b | Phase 2
Started | 9 | 0
Completed | 7 | 0
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Population: The study was terminated after the Phase 1b completed and prior to Phase 2 initiation.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1b | Phase 2 | Total
Number analyzed (Participants) | 9 | 0 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 0 | 6
  >=65 years | 3 | 0 | 3
Age, Continuous [Mean (Full Range); unit: years] | 62.3 [52 to 70] |  | 62.3 [52 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 0 | 4
  Male | 5 | 0 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 8 | 0 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 0 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 |  | 9

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Determine the clinical activity as defined by overall response rate (ORR) of bemcentinib plus chemotherapy (nab-paclitaxel/gemcitabine) in patients with metastatic pancreatic adenocarcinoma. The analyses of ORR was performed on the Response Evaluable Population. ORR is defined as the proportion of patients with CR+partial response as their best clinical response.
Time Frame: Every 4 months from time of first dose of study drug until completion of treatment for approximately 42 months.
Population: The study was terminated after the Phase 1b completed and prior to Phase 2 initiation.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b | Phase 2
Number analyzed (Participants) | 7 | 0
Participants | 2 | 0

2. Secondary Outcome: Complete Response Rate (CR)
Description: Determine clinical activity of bemcentinib plus chemotherapy as defined by complete response rate (CRR), partial response, stable disease, duration of response - overall response/stable disease, median progression free survival (PFS) and overall survival (OS) rate.
Time Frame: Every 4 months from time of first dose of study drug until completion of treatment for approximately 42 months.
Population: The study was terminated after the Phase 1b completed and prior to Phase 2 initiation.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b | Phase 2
Number analyzed (Participants) | 7 | 0
Participants | 0 | 0

3. Secondary Outcome: Clinical Benefit Rate
Description: Determine clinical benefit rate as defined by complete response (CR), Partial Response (PR), and Stable Disease (SD) response rates. Clinical benefit response - percent of CR, PR, and SD.
Time Frame: Every 4 months from time of first dose of study drug until completion of treatment for approximately 42 months.
Population: The study was terminated after the Phase 1b completed and prior to Phase 2 initiation.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b | Phase 2
Number analyzed (Participants) | 7 | 0
Participants | 6 | 0

4. Secondary Outcome: Number of Participants With an Adverse Event of Grade 3 or Higher
Description: Assess safety and tolerability of bemcentinib plus chemotherapy in patients with metastatic pancreatic adenocarcinoma and will be graded according to the NCI CTCAE, Version 5
Time Frame: Every 4 months from time of first dose of study drug until completion of treatment for approximately 42 months.
Population: 5 patients experienced an adverse event of grade 3 or higher. The study was terminated after the Phase 1b completed and prior to Phase 2 initiation.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b | Phase 2
Number analyzed (Participants) | 9 | 0
Participants | 5 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over a time period of approximately 42 months.
Description: The study was terminated after the Phase 1b completed and prior to Phase 2 initiation.
Arm/Group | Phase 1b | Phase 2
All-Cause Mortality (participants affected / at risk) | 1/9 | 0/0
Serious Adverse Events (participants affected / at risk) | 4/9 | 0/0
Other Adverse Events (participants affected / at risk) | 9/9 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1b (N=9) | Phase 2 (N=0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Allergic Reaction (Immune system disorders) | 1 (1) | NA
Diarrhea (Gastrointestinal disorders) | 1 (1) | NA
Sepsis (Infections and infestations) | 2 (2) | NA
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | NA
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | NA
Localized Edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA
Anemia (Blood and lymphatic system disorders) | 1 (1) | NA
Urine Discoloration (Immune system disorders) | 1 (1) | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1b (N=9) | Phase 2 (N=0)
Anemia (Blood and lymphatic system disorders) | 4 (20) | NA
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | NA
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | NA
Alkaline Phosphatase Increased (Hepatobiliary disorders) | 1 (2) | NA
Anorexia (Metabolism and nutrition disorders) | 2 (2) | NA
Allergic Reaction (Immune system disorders) | 1 (5) | NA
Ascites (Gastrointestinal disorders) | 1 (2) | NA
Creatinine Increased (Renal and urinary disorders) | 2 (3) | NA
Constipation (Gastrointestinal disorders) | 3 (3) | NA
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA
Dizziness (Nervous system disorders) | 2 (2) | NA
Diarrhea (Gastrointestinal disorders) | 4 (5) | NA
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (5) | NA
Dysgeusia (Nervous system disorders) | 1 (1) | NA
Dysphagia (Gastrointestinal disorders) | 1 (1) | NA
ECG QT corrected interval prolonged (Cardiac disorders) | 1 (1) | NA
Fatigue (General disorders) | 7 (8) | NA
Fever (General disorders) | 1 (1) | NA
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA
GERD (Gastrointestinal disorders) | 4 (4) | NA
Hypokalemia (Metabolism and nutrition disorders) | 2 (4) | NA
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (5) | NA
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | NA
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (3) | NA
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | NA
Hyponatremia (Investigations) | 1 (2) | NA
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | NA
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | NA
Nausea (Gastrointestinal disorders) | 6 (6) | NA
Localized Edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA
Neutrophil Count Decreased (Blood and lymphatic system disorders) | 4 (6) | NA
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | NA
Mucositis Oral (Infections and infestations) | 1 (1) | NA
Lymphocyte Count Decreased (Blood and lymphatic system disorders) | 3 (3) | NA
Pain (Gastrointestinal disorders) | 4 (4) | NA
Peripheral Sensory Neuropathy (Nervous system disorders) | 4 (4) | NA
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA
Pulmonary Embolism (Vascular disorders) | 1 (1) | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (4) | NA
Sepsis (Infections and infestations) | 2 (2) | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (11) | NA
Thrush (Infections and infestations) | 1 (1) | NA
Tumor Lysis Syndrome (Metabolism and nutrition disorders) | 1 (1) | NA
Tinnitus (Ear and labyrinth disorders) | 1 (1) | NA
Vomiting (Gastrointestinal disorders) | 3 (4) | NA
Upper Respiratory Infection (Infections and infestations) | 1 (1) | NA
Urine Discoloration (Renal and urinary disorders) | 2 (2) | NA
WBC Count Decreased (Blood and lymphatic system disorders) | 1 (1) | NA
Skin Infection (Skin and subcutaneous tissue disorders) | 1 (2) | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-01): https://cdn.clinicaltrials.gov/large-docs/21/NCT03649321/Prot_SAP_000.pdf
  • Informed Consent Form (2021-08-09): https://cdn.clinicaltrials.gov/large-docs/21/NCT03649321/ICF_001.pdf